CLINICAL TRIAL: NCT01497808
Title: RADVAX™: A STRATIFIED PHASE I/II DOSE ESCALATION TRIAL OF HYPOFRACTIONATED RADIOTHERAPY FOLLOWED BY IPILIMUMAB IN METASTATIC MELANOMA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06611
Record Dates: First submitted 2011-12-13; First posted 2011-12-23 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Melanoma
Keywords: previously untreated; previously treated; bone, lung, liver or subcutaneous involvement; nodal involvement; without evidence of brain involvement
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ipilimumab and Radiotherapy (8 Gy x 2) (Experimental)
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy
- Ipilimumab and Radiotherapy (8 Gy x 3) (Experimental)
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy
- Ipilimumab and Radiotherapy (6 Gy x 2) (Experimental)
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy
- Ipilimumab and Radiotherapy (6 Gy x 3) (Experimental)
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Ipilimumab
Radiation: Stereotactic Body Radiation Therapy

SUMMARY:
The primary objective is to determine the maximum tolerated hypofractionated radiotherapy dose (MTD) to a solitary metastatic focus ('index lesion') when followed by ipilimumab, in metastatic melanoma patients without brain involvement The secondary objectives are to determine late toxicity, immune-related clinical responses and immune pharmacodynamic changes after hypofractionated radiotherapy followed by ipilimumab

ELIGIBILITY:
Inclusion Criteria

* Patient > 18 years old
* Histologically confirmed diagnosis of melanoma
* Previously treated or previously untreated metastatic melanoma by AJCC staging criteria
* Presence of an index lesion > 1 cm amenable to hypofractionated radiotherapy and at least one other additional lesion that can be followed for response using RECIST criteria
* ECOG Performance status 0 or 1
* Signed informed consent document
* Ability to tolerate stereotactic body radiation therapy (e.g. lie flat and hold position for treatment)

Exclusion Criteria

* Prior systemic therapy within 14 days of study enrollment. Patients must be adequately recovered from prior systemic therapy side effects as deemed by the PI.
* Clinical contraindication to stereotactic body radiotherapy (e.g. active systemic sclerosis, active inflammatory bowel disease if bowel is within target field, etc)
* Presence or history of central nervous system metastasis (including brain)
* Long-term use of systemic corticosteroids
* Prior RT that precludes the delivery of hypofractionated radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2013-12-29 (Actual); Study Completion 2015-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Maity, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the Universirty of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Maity A, Mick R, Rengan R, Mitchell TC, Amaravadi RK, Schuchter LM, Pryma DA, Patsch DM, Maity AP, Minn AJ, Vonderheide RH, Lukens JN. A stratified phase I dose escalation trial of hypofractionated radiotherapy followed by ipilimumab in metastatic melanoma: long-term follow-up and final outcomes. Oncoimmunology. 2021 Jan 31;10(1):1863631. doi: 10.1080/2162402X.2020.1863631. PMID 33643689

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab and Radiotherapy (8 Gy x 2): Ipilimumab
  Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | Ipilimumab and Radiotherapy (8 Gy x 2) | Ipilimumab and Radiotherapy (8 Gy x 3) | Ipilimumab and Radiotherapy (6 Gy x 2) | Ipilimumab and Radiotherapy (6 Gy x 3)
Started | 6 | 4 | 6 | 6
Completed | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab and Radiotherapy (8 Gy x 2) | Ipilimumab and Radiotherapy (8 Gy x 3) | Ipilimumab and Radiotherapy (6 Gy x 2) | Ipilimumab and Radiotherapy (6 Gy x 3) | Total
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 0 | 8
  >=65 years | 3 | 1 | 4 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 5
  Male | 5 | 2 | 5 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 6 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 6 | 6 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab and Radiotherapy (8 Gy x 2) | Ipilimumab and Radiotherapy (8 Gy x 3) | Ipilimumab and Radiotherapy (6 Gy x 2) | Ipilimumab and Radiotherapy (6 Gy x 3)
Number analyzed (Participants) | 6 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Participants With Adverse Events
Time Frame: after 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab and Radiotherapy (8 Gy x 2) | Ipilimumab and Radiotherapy (8 Gy x 3) | Ipilimumab and Radiotherapy (6 Gy x 2) | Ipilimumab and Radiotherapy (6 Gy x 3)
Number analyzed (Participants) | 6 | 4 | 6 | 6
Participants | 6 | 4 | 6 | 6

ADVERSE EVENTS:
Arm/Group | Ipilimumab and Radiotherapy (8 Gy x 2) | Ipilimumab and Radiotherapy (8 Gy x 3) | Ipilimumab and Radiotherapy (6 Gy x 2) | Ipilimumab and Radiotherapy (6 Gy x 3)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/6 | 1/4 | 3/6 | 2/6
Other Adverse Events (participants affected / at risk) | 5/6 | 3/4 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab and Radiotherapy (8 Gy x 2) (N=6) | Ipilimumab and Radiotherapy (8 Gy x 3) (N=4) | Ipilimumab and Radiotherapy (6 Gy x 2) (N=6) | Ipilimumab and Radiotherapy (6 Gy x 3) (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
(General disorders) | 4 | 1 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab and Radiotherapy (8 Gy x 2) (N=6) | Ipilimumab and Radiotherapy (8 Gy x 3) (N=4) | Ipilimumab and Radiotherapy (6 Gy x 2) (N=6) | Ipilimumab and Radiotherapy (6 Gy x 3) (N=6)
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
(General disorders) | 4 | 3 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes